CLINICAL TRIAL: NCT01716429
Title: Healthy Eating for Reproductive Health: Greenville
Acronym: HER Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were recruited over the course of the study time period
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019109
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2013-09

CONDITIONS: Polycystic Ovarian Syndrome; Infertility; Obesity; Overweight
Keywords: vegetarian; vegan; low calorie; weight Loss; infertility; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Obesity; Overweight; Weight Loss | interventions — Diet, Vegan; Diet, Vegetarian; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Calorie (Active Comparator): Participants in this arm will be instructed on how to reduce their caloric intake and follow a low calorie diet
  Interventions: Behavioral: Low calorie diet
- Vegan diet (Experimental): Participants in this arm will follow a very low fat diet (~10% kcals from fat) and also a diet that has a low glycemic index and is free of animal products (vegan)
  Interventions: Behavioral: Vegan diet

INTERVENTIONS:
Behavioral: Vegan diet — Vegan dietary approaches for weight loss
  Other Names: Vegetarian
  Arms: Vegan diet
Behavioral: Low calorie diet — Reduced calorie diet for weight loss
  Other Names: Standard diet
  Arms: Low Calorie

SUMMARY:
This study will be a 6-month intervention that is examining how different dietary approached may be useful for women with Polycystic Ovarian Syndrome (PCOS) who are attempting pregnancy, particularly by measuring changes in weight. Participants will be randomly assigned to following one of two dietary approaches for weight loss: 1) a low-calorie approach to weight loss (reducing caloric intake by approximately 500 calories per day) or 2) a low-fat, low-glycemic index vegan diet. A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. In addition, this diet will be low-glycemic index, which means the consumer will be asked to favor foods that don't cause a quick rise in blood sugar (for example, favoring oatmeal over cornflakes for breakfast). Participants will receive counseling and supporting materials on the dietary approach the participants are assigned to follow. Both diets are safe and have shown to be effective ways to assist with achieving a healthy weight. The investigators hypothesize that both groups will see improvements in weight and fertility with possible greater improvements seen among participants in the vegan group.

DETAILED DESCRIPTION:
This study involves two groups. You will be randomly assigned to one of these groups (i.e. you do not have a choice for group assignment) which means your group will be assigned to you by chance. Both groups will receive information on a dietary approach aimed at losing weight.

One group will receive instruction on a low-calorie approach to weight loss (reducing caloric intake by approximately 500 calories per day). The other group will be instructed to follow a low-fat, low-glycemic index vegan diet. A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. In addition, this will be a low-glycemic index diet, which means you will be asked to favor foods that don't cause a quick rise in blood sugar (for example, choosing oatmeal over cornflakes for breakfast).

Below are the steps in the study:

If you are accepted into the study, you will come to the study site (Fertility Center of the Carolinas in Greenville) to learn more about the study and complete your consent form. If you live outside the Columbia, SC area (more than a 60 mile drive), you may complete the study orientation process over the phone and Web. You will be mailed a consent form to sign and return to the study coordinator. This study will involve 3-4 in-person visits to the Fertility Center of the Carolinas office, each lasting approximately 1.5 to 2 hours.

You will complete some questionnaires that measure your diet and physical activity levels on a computer at home or other location where you have computer/internet access.

You will come back for a meeting to have your weight measured. You will then be randomly assigned to one of the two groups: calorie controlled group or vegan diet group. You will receive a one-hour overview of the diet you have been assigned to and be provided with materials on this diet.

During the study, we will ask you to complete a weekly questionnaire which will assess if you are following the diet, your weight, and ask for information on your menstrual cycle. This will take approximately 5 minutes to complete.

You will be provided individualized feedback each week via e-mail on your progress, along with a weekly lesson on the topic for the week.

You will have access to a group website (a private Facebook group) that will provide group support. Participation using this group is optional.

You will be provided with test strips to monitor ovulation each month and pregnancy tests (1 per month) to monitor pregnancy status. You will report these results to us via online survey.

Study personnel will host a weekly 30 minute webinar for your diet group online. This will take place after work time on a weekday. Make-up sessions by phone during the work day will be available.

At 3 months, you will be asked to complete another set of questionnaires from home and return to our study site for your weight measurement.

You will continue the study for the next 3 months. At study completion (6 months), you will complete the last set of questionnaires (online). Also, you will come to a follow-up assessment to be weighed and to receive your incentive for participating ($10 +$5/month of each menstrual cycle data submitted for a total of $25 possible).

Participants in both groups will be asked to take a daily prenatal vitamin (or other reliable source of vitamin B-12) over the course of the study.

During the study, we will ask you to keep your physical activity levels constant (keep your levels the same as what you were doing at study entry).

ELIGIBILITY:
Inclusion Criteria:

Women must meet the following criteria:

have been attempting pregnancy for at least 6 months is not currently pregnant has a clinical diagnosis of PCOS is not on oral medications for insulin resistance (such as metformin) or, if currently on such a medication, has been on the medication at a stable dose for at least 3 months willing not use fertility-enhancing medications over the 6-month study (with the exception of oral medications, such as clomiphene citrate, as directed by their physician) willing to be randomized to either dietary condition and able to make weekly meetings.

Exclusion Criteria:

Participants should not be in this study if they meet any of the following criteria:

have not been diagnoses with polycystic ovarian syndrome have been trying to conceive less than 6 months have a Body Mass Index less than 25 or greater than 45 kg/m2 are currently pregnant are younger than 18 or older than 35 years of age are a smoker are unable to come to the Columbia, SC area at least 3-4 times in a 6 month time period for assessments don't have access to the Internet and a computer don't have access to a scale for self-monitoring weight aren't willing to be randomized to either group have a psychiatric disease, drug or alcohol dependency, or uncontrolled thyroid condition have a major health condition, such as heart conditions, diabetes, and past incidence of stroke unable to receive consent from your doctor to participate if you currently are on blood pressure medications, have issues with dizziness, or have bone or joint issues have an eating disorder currently participating in a weight loss program or taking weight loss medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | 6 months

SECONDARY OUTCOMES:
Pregnancy rates | 6 months

OTHER OUTCOMES:
Menstrual cycle length | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Fertility Center of the Carolinas: Greenville Hospital System, Greenville, South Carolina, United States